CLINICAL TRIAL: NCT06595576
Title: Dose-dependent Effects of Cannabis Edibles on Simulated Driving Performance
Brief Title: Cannabis Edibles and Simulated Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 074-2020
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-02

CONDITIONS: Cannabis; Driving Under the Influence
Keywords: Cannabis Edibles; THC; Driving Simulator; Cognition; Subjective Effects; Cannabinoids
MeSH Terms: conditions — Marijuana Abuse; Driving Under the Influence | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: The study will be a within-subjects, double-blind, placebo-controlled, randomized and counterbalanced human laboratory experiment assessing the effects of a range of doses of cannabis edibles on driving simulator performance. These 4 drug exposure conditions are: placebo, low dose (2 + 2% mg THC), medium dose (10 + 2% mg THC), and high dose (20 + 2% mg THC).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo Cannabis Edibles (0 mg THC) (Experimental): Participants consume a placebo dose of cannabis edibles (0 mg THC).
  Interventions: Drug: Cannabis - Placebo Dose (0 mg)
- Low Dose Cannabis Edibles (2 mg THC) (Experimental): Participants consume a low dose of cannabis edibles (2 mg THC).
  Interventions: Drug: Cannabis - Low Dose (2 mg)
- Medium Dose Cannabis Edibles (10 mg) (Experimental): Participants consume a medium dose of cannabis edibles (10 mg THC).
  Interventions: Drug: Cannabis - Medium Dose (10 mg)
- High Dose Cannabis Edibles (20 mg) (Experimental): Participants consume a high dose of cannabis edibles (20 mg THC).
  Interventions: Drug: Cannabis - High Dose (20 mg)

INTERVENTIONS:
Drug: Cannabis - Placebo Dose (0 mg) — Participants will consume placebo cannabis edibles.
  Arms: Placebo Cannabis Edibles (0 mg THC)
Drug: Cannabis - Low Dose (2 mg) — Participants will consume a low dose (2 mg) of cannabis edibles.
  Arms: Low Dose Cannabis Edibles (2 mg THC)
Drug: Cannabis - Medium Dose (10 mg) — Participants will consume a medium dose (10 mg) of cannabis edibles.
  Arms: Medium Dose Cannabis Edibles (10 mg)
Drug: Cannabis - High Dose (20 mg) — Participants will consume a high dose (20 mg) of cannabis edibles.
  Arms: High Dose Cannabis Edibles (20 mg)

SUMMARY:
The goal of this human laboratory experiment is to determine the acute and residual effects of a range of doses of orally administered cannabis edibles on driving simulator performance in people who use cannabis recreationally. Four conditions will be tested: placebo, low dose, medium dose and high dose. Driving performance will be tested objectively using a driving simulator during a number of pre-programmed driving scenarios. The investigators will test the hypothesis that driving performance on a high-fidelity driving simulator will decrease with increasing doses of cannabis. Secondary objectives will:

* Determine the acute and residual (24 hour) cognitive, behavioural, and physiological effects of a range of doses of orally administered cannabis edibles on subjective effects, cognitive tests, verbal memory, and mood.
* Examine how the concentration of THC in blood and oral fluids correlates with driving simulator performance, as well as cognitive, behavioural, and physiological measures. Cannabinoid levels in blood, urine and oral fluids will be measured at baseline and over a 5 hour period following drug exposure. The investigators will examine the relationship between cannabinoid levels and performance measures in this time frame.
* Explore potential biomarkers of acute exposure to cannabis edibles by analyzing the following: circulating cell-free mtDNA (ccf-mtDNA), endocannabinoids, and metabolic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Provides written and informed consent
* Stated the willingness to comply with all study procedures
* Recreational use of oral, vaped, smoked or edible cannabis (at least one day/week) and cannabis edibles (at least one day/month) confirmed by self-report and urine screening (i.e., positive THC result in point-of-care screening or Clinical Laboratory assay)
* Males and females aged 19 to 45 years
* Has held a class G license (or equivalent from another jurisdiction) for at least 12 months
* Willing to abstain from using cannabis for 72 hours prior to each practice or test session
* Willing to abstain from alcohol for 48 hours prior to each practice or test session, and to abstain from all other drugs not medically required for the duration of the study (beginning 48 hours prior to the practice session)
* Lives within a radius that costs less than about $60 per taxi ride
* Able to consume the quantity of candies and drive the driving simulator as determined by a practice session
* A negative urine pregnancy test for those with childbearing potential
* Use of appropriate contraception for those with childbearing potential

Exclusion Criteria:

* Diagnosis of severe medical or psychiatric condition (e.g., diagnosis of a severe mood or anxiety disorder, based on self-report
* Meets criteria for current or lifetime alcohol or other substance use disorder (DSM-5), except tobacco use disorder and caffeine use disorder
* Regular user of medication that may affect cognitive functioning and/or driver performance (e.g. ADHD medication, benzodiazepines, stimulants, opioids)
* Regular user of illicit substances
* Personal or family history of schizophrenia or other psychotic disorder
* Pregnant, looking to become pregnant, or breastfeeding
* Concomitant therapy with sedative-hypnotics or other psychoactive drugs
* Severe laboratory abnormalities that could create safety issues based on the judgement of the Principal Investigator
* Cardiovascular or cerebrovascular disease
* Severe renal or liver disease
* Participation in another clinical or non-therapeutic study in the past month

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Standard Deviation of Lateral Position (SDLP) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  The driving simulator will objectively record SDLP during a number of pre-programmed driving scenarios.

SECONDARY OUTCOMES:
Mean Speed (MS) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  The driving simulator will objectively record MS during a number of pre-programmed driving scenarios.
Reaction Time (RT) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  The driving simulator will objectively record RT during a number of pre-programmed driving scenarios.
Standard Deviation of Speed (SDS) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  The driving simulator will objectively record SDS during a number of pre-programmed driving scenarios.
Blood concentrations of Δ9-tetrahydrocannabinol (THC), 11-hydroxy-Δ9-tetrahydrocannabinol (OH-THC), and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol (THC-COOH) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess THC and metabolite concentrations (ng/mL) in blood.
Oral fluid concentrations of Δ9-tetrahydrocannabinol (THC), 11-hydroxy-Δ9-tetrahydrocannabinol (OH-THC), and 11-Nor-9-carboxy-Δ9-tetrahydrocannabinol (THC-COOH) and point-of-care detection of cannabinoids | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess THC and metabolite concentrations (ng/mL) in oral fluid.
Heart Rate | Before cannabis exposure; 0, 30, 60, 90 minutes and 2, 3, 4 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated approximately 24 hours after dosing.
  Heart rate (bpm) will be measured.
Blood Pressure | Before cannabis exposure; 0, 30, 60, 90 minutes and 2, 3, 4 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated approximately 24 hours after dosing.
  Systolic and diastolic blood pressure (mmHg) will be measured.
Temperature | Before cannabis exposure; 0, 30, 60, 90 minutes and 2, 3, 4 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated approximately 24 hours after dosing.
  Temperature (degrees Celsius) will be measured.
Visual Analog Scale (VAS) | Before cannabis exposure; 0, 30, 60, 90 minutes and 2, 3, 4 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated approximately 24 hours after dosing.
  Used to assess subjective effects of cannabis on a sliding scale of 0 (not at all) to 100 (maximum effect).
Addiction Research Centre Inventory (ARCI) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess subjective effects of cannabis.
Profile of Mood States (POMS) | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess subjective effects of cannabis.
Verbal Free Recall Task | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess the impact of cannabis on verbal learning and memory.
Blood Concentrations of mtDNA | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess concentrations of mtDNA.
Blood Concentrations Endocannabinoids | Before cannabis exposure; 2 and 5 hours after cannabis exposure (repeated each session for 4 sessions). Also repeated on the test for residual effects, approximately 24 hours after dosing.
  Used to assess concentrations of endocannabinoids.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada